CLINICAL TRIAL: NCT06405490
Title: Nanoliposomal Irinotecan and XELOX (NALIRI-XELOX) in Combination With Cadonilimab for First-Line Treatment of Patients With Locally Advanced or Metastatic Pancreatic Ductal Adenocarcinoma : A Single-arm, Phase II Study
Brief Title: NALIRI-XELOX+AK104 for First-line Treatment of Advanced PDAC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, LIN YANG, chief physician, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC4398
Record Dates: First submitted 2024-05-05; First posted 2024-05-08 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Nanoliposomal Irinotecan; Cadonilimab; Oxaliplatin; Capecitabine; First-Line; Advanced Cancer; Pancreatic Adenocarcinoma; Drug Use
Keywords: Pancreatic Adenocarcinoma; Nanoliposomal Irinotecan; Cadonilimab; First-Line Treatment; Advanced Pancreatic Adenocarcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NALIRI-XELOX+AK104 (Experimental): Every 2 weeks as a cycle:
  1. Nanoliposomal Irinotecan: 47.1mg/m2, iv, d1;
  2. Cadonilimab: 6mg/kg, iv, d3;
  3. Oxaliplatin: 70mg/m2, iv, d1;
  4. Capecitabine: 1000mg/m2, bid, po, d1-d7; Re-evaluate patients every three cycles. If the patient has been treated for more than 9 cycles, they will enter maintenance therapy, and the regimen is capecitabine +Cadonilimab.
  Interventions: Drug: Nanoliposomal Irinotecan+Oxaliplatin +Capecitabine+Cadonilimab

INTERVENTIONS:
Drug: Nanoliposomal Irinotecan+Oxaliplatin +Capecitabine+Cadonilimab — Use the above medications on a regular basis

SUMMARY:
This study is a single-center, Phase II Study to assess the efficacy and safety of the regimen of Nanoliposomal Irinotecan and XELOX (NALIRI-XELOX) in combination with Cadonilimab in subjects with advanced pancreatic ductal adenocarcinoma who have not previously received systemic treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18, male or female;
2. Has histologically or cytologically confirmed pancreatic ductal adenocarcinoma (PDAC);
3. Has not received prior systemic treatment for their locally advanced or metastatic PDAC;
4. Has presence of measurable disease as defined by Response Evaluation Criteria in Solid Tumours (RECIST 1.1);
5. Has a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Status;
6. Has a life expectancy of at least 3 months;
7. Has adequate organ function;
8. If female of childbearing potential, have a negative serum pregnancy test within 7 days prior to first trial treatment;
9. If female of childbearing potential or a male subject with a partner with childbearing potential, be willing to use a highly effective method of contraception (with a failure rate of less than 1.0% per year) from first study treatment to 24 weeks after completion of the trial treatment.

Exclusion Criteria:

1. Untreated active CNS metastasis or leptomeningeal metastasis.
2. Is currently participating and receiving an investigational drug or has participated in a study of an investigational drug within 4 weeks or within 5 times of half-life (no less than 2 weeks), whichever is shorter prior to the first dose of trial treatment;
3. Has received other anti-tumor treatment within 4 weeks or within 5 times of half-life (no less than 2 weeks), whichever is shorter prior to the first trial treatment;
4. Major surgery for any reason, except diagnostic biopsy, within 4 weeks of the first administration of trial treatment and/or if the subject has not fully recovered from the surgery within 4 weeks of the first administration of trial treatment;
5. Curative radiation within 3 months of the first dose of trial treatment. Radiation to more than 30% of the bone marrow or with a wide field of radiation should not be used within 4 weeks prior to the first administration of trial treatment;
6. Subjects receiving immunosuppressive agents (such as steroids) for any reason should be tapered off these drugs before initiation of trial treatment (with the exception of subjects with adrenal insufficiency, who may continue corticosteroids at physiologic replacement doses, equivalent to < 10 mg prednisone daily, inhaled steroids and topical use of steroids);
7. Vaccination within 28 days of the first administration of trial treatment, except for administration of inactivated vaccines (e.g., inactivated influenza vaccines);
8. Has interstitial lung disease, or a history of pneumonitis that required oral or intravenous glucocorticoids to assist with management;
9. History or current active autoimmune disease that might deteriorate when receiving an immunostimulatory agent；
10. Previous malignant disease History of uncontrolled intercurrent illness Prior therapy with any antibody/drug targeting T cell coregulatory proteins Known severe hypersensitivity reactions to antibody drug；
11. Is pregnant or breastfeeding;
12. Other medical conditions that at the discretion of investigator interfere with the requirements of the trial in terms of safety or efficacy evaluation, or treatment compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 2 years
  ORR of regimen of NALIRI-XELOX+AK104

SECONDARY OUTCOMES:
Duration of Response (DoR) | 2 years
Disease Control Rate (DCR) | 2 years
Median Progression-Free Survival (mPFS) | 1 years
12-month PFS rate | 12 months
Median Overall Survival (mOS) | 2 years
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] Adverse Events (AEs) Incidence, Serious Adverse Events (SAE) Incidence | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China